CLINICAL TRIAL: NCT01283256
Title: Evaluation of Safety and Efficacy of Zonisamide in Adult Patients With Partial, Generalized and Combined Seizures: An Open Labeled, Non-comparative, Observational Study
Brief Title: A Study to Evaluate the Safety and Efficacy of Zonisamide an Antiepileptic Drug as Monotherapy or Adjunctive Therapy in Treatment of Adult Patients With Partial, Generalized or Combined Seizures.
Status: Completed | Type: Observational
Sponsor: Eisai Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: EIL/ZONE/CT01/2010
Record Dates: First submitted 2011-01-24; First posted 2011-01-25 (Estimated); Last update posted 2014-01-27 (Estimated); Status verified 2014-01

CONDITIONS: Partial, Generalized and Combined Seizures
MeSH Terms: interventions — Zonisamide

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (1):
- Experimental
  Interventions: Drug: zonisamide

INTERVENTIONS:
Drug: zonisamide — zonisamide 100mg tablets

SUMMARY:
The purpose of this study is to evaluate the safety and efficacy of zonisamide in the treatment of adult patients with partial, generalized or combined seizures.

DETAILED DESCRIPTION:
This is an open labeled non-comparative, multicentric observational post marketing surveillance study to comparing the safety and efficacy of zonisamide as adjunctive therapy or monotherapy in patients with partial, generalized or combined seizures, in a initiating dose of 100mg/day titrated to a maximum of 600mg per day based on the seizure control and tolerability over a 24 weeks treatment period. This study will include a total of 900 patients with partial, generalized or combined seizures across 30 centres in the country. The patients will be enrolled based on the inclusion and exclusion criteria and will be evaluated for safety and efficacy at every 4 weekly interval for 24 weeks. There will be total 7 study visits and the patients will be evaluated for clinically reportable adverse events, safety on Patients Global Assessment of Tolerability to Therapy (PGATT) on a 4-point scale and for efficacy by evaluation of reduction in seizure frequency as the primary objective of the study. For secondary objectives the patients data will be evaluated to determine the responder rates (> or = to 50% reduction in seizure frequency from baseline) and seizure freedom over the 24 weeks study period.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female subjects, 18 to 75 years of age inclusive
2. Treated or untreated subjects suffering from any of the following types of seizures:

   1. Partial Seizures: Simple Partial Seizures, Complex Partial Seizures & Secondarily generalized tonic clonic seizures
   2. Generalized Seizures: Tonic-clonic seizures, tonic seizures & Atypical absence seizures
   3. Combined seizures (mixed)
3. Subjects having had a computed tomography (CT) or magnetic resonance imaging (MRI) done within the last upto 10 years that ruled a progressive cause of epilepsy.
4. Female subjects without child bearing potential (2 years postmenopausal, bilateral oophorectomy or tubal ligation, complete hysterectomy) are eligible.
5. Female subjects with childbearing potential must not be pregnant as confirmed by a negative pregnancy test at screening and enrollment must not be lactating and must be using a medically acceptable form of contraception, for the duration of the study and for one month following discontinuation of the study drug.
6. Patients willing to take the medications as directed, maintain a seizure dairy, report adverse events and willing to come for the follow-ups as per schedule.
7. Willing to comply with the protocol requirements.
8. Able and willing to give the written informed consent.

Exclusion Criteria:

1. Subjects with history of non-epileptic seizures (e.g. metabolic, pseudo-seizures).
2. Subjects who have experienced seizures relating to drugs, alcohol, acute medical illness, mental retardation, or subjects with situation related seizures.
3. Subjects with progressive encephalopathy or findings consistent with progressive CNS disease or lesion (e.g. infection, demyelination or tumour).
4. Subjects with a history of any significant or currently uncontrolled disease which in the opinion of the investigator will interfere with the conduct of this study or the assessment of safety & efficacy of the study drug.
5. Subjects already receiving zonisamide therapy.
6. Subjects who have received an investigational new drug or device in the past three months before screening and enrollment.
7. Subjects with known hypersensitivity to zonisamide or sulphonamides.
8. Subjects with known abnormal renal function (serum creatinine > 1.5 mg/dL) or abnormal hepatic function (Aspartate aminotransferase [AST] and alanine aminotransferase [ALT] > 2 times the upper normal limit).
9. Subjects with a history of psychiatric illness or mood disorder requiring electro-convulsive or drug therapy within previous 6 months which is considered uncontrolled; a history of suicide attempt; alcohol or drug abuse.
10. Subjects currently taking carbonic anhydrase inhibitors (acetazolamide).
11. Subjects currently taking Mono-Amine Oxidase Inhibitor's (MAO-I's).
12. Subjects having a history of pancreatitis, nephrolithiasis or hypercalciuria, clinically significant laboratory abnormalities suggestive of metabolic imbalance

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Single Cohort Study involving community patients with epilepsy
Sampling Method: Non-Probability Sample
Enrollment: 655 (Actual)
Dates: Start 2011-01; Primary Completion 2013-01 (Actual); Study Completion 2013-05 (Actual)

PRIMARY OUTCOMES:
Assess safety with zonisamide therapy in adult patients with different seizure types | 24 weeks
Assess reduction in seizure frequency with zonisamide therapy in adult patients with different seizure types | 24 weeks

SECONDARY OUTCOMES:
To evaluate responder rates over 24 weeks of zonisamide treatment in adult patient with seizures | 24 weeks
To evaluate seizure freedom over 24 weeks of zonisamide treatment in adult patient with seizures | 24 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Amitabh Dash, Study Director — Eisai Pharmaceuticals India Private limited
Locations (14):
- India (14):
  - Hyderabad, Andhra Pradesh
  - Secunderabad, Andhra Pradesh
  - Vijaywada, Andhra Pradesh
  - Visakhapatnam, Andhra Pradesh
  - Ahmedabad, Gujarat
  - Bangalore, Karnataka
  - Kochi, Kerala
  - Mumbai, Maharashtra
  - Pune, Maharashtra
  - New Delhi, New Delhi
  - Jaipur, Rajasthan
  - Chennai, Tamil Nadu
  - Lucknow, Uttar Pradesh
  - Noida, Uttar Pradesh